CLINICAL TRIAL: NCT04557605
Title: The Effects of Wearing a Face Mask During COVID-19 on Blood and Muscle Oxygenation While Performing Exercise
Brief Title: Effects of a Face Mask on Oxygenation During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2201
Record Dates: First submitted 2020-09-09; First posted 2020-09-21 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The individual who will statistically analyze the data will be blinded to condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No face mask (Active Comparator): Progressive step-exercise cycling test to exhaustion wearing no face mask
  Interventions: Other: Progressive cycling exercise test to exhaustion
- Disposable face mask (Experimental): Progressive step-exercise cycling test to exhaustion wearing a 3-ply disposable face mask
  Interventions: Other: Progressive cycling exercise test to exhaustion
- Cloth face mask (Experimental): Progressive step-exercise cycling test to exhaustion wearing a cloth face mask
  Interventions: Other: Progressive cycling exercise test to exhaustion

INTERVENTIONS:
Other: Progressive cycling exercise test to exhaustion — Progressive step cycling exercise test to exhaustion

SUMMARY:
There is concern that wearing a face mask during COVID will affect oxygen uptake, especially during intense exercise. This study will assess the effect of wearing two different face masks (disposable and cloth) on blood and muscle oxygenation during cycling exercise.

DETAILED DESCRIPTION:
There is concern that wearing a face mask during exercise will reduce oxygen uptake or increase carbon dioxide re-breathing, which can result in low blood oxygen levels, reduced oxygen delivery to muscle and reduced exercise capacity. The purpose of the study is to determine the effect of wearing two different types of commonly-worn face masks (diposable and cloth) during exercise on blood and muscle oxygenation. Twelve participants who are experienced with cycling will take part in this randomized cross-over study that will assess blood oxygenation (i.e. pulse oximetry) and muscle oxygenation (with near infrared spectroscopy) during a progressive step exercise test to exhaustion. The conditions include no mask, a disposable mask, and a cloth mask. Outcome variables include exercise duration, rating of perceived exertion, blood oxygen saturation levels, and oxygenated, deoxygenated, and total hemoglobin at the quadriceps muscle.

ELIGIBILITY:
Inclusion Criteria:

* Experienced with cycling

Exclusion Criteria:

* Contra-indications to exercise as identified by a screening questionnaire (the "Get Active Questionnaire")

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Time to exhaustion during exercise | Up to 20 minutes
  time to exhaustion
Change from baseline in peak power output | Up to 20 minutes
  Peak power output in Watts, determined on a cycle ergometer

SECONDARY OUTCOMES:
Change from baseline in blood oxygen saturation | Up to 20 minutes
  Blood oxygen saturation as determined by pulse oximetry
Change from baseline in quadriceps tissue oxygenation index | Up to 20 minutes
  Tissue oxygenation index (oxygenated hemoglobin/total hemoglobin) as measured by near infra-red spectroscopy
Change from baseline in rating of perceived exertion | Up to 20 minutes
  Rating of perceived exertion on a scale of 1-10 (Modified Borg Scale), a higher score indicates a greater perceived exertion
Change from baseline in heart rate | Up to 20 minutes
  Heart rate (beats per minute)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chilibeck, Ph.D., Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shaw K, Butcher S, Ko J, Zello GA, Chilibeck PD. Wearing of Cloth or Disposable Surgical Face Masks has no Effect on Vigorous Exercise Performance in Healthy Individuals. Int J Environ Res Public Health. 2020 Nov 3;17(21):8110. doi: 10.3390/ijerph17218110. PMID 33153145